CLINICAL TRIAL: NCT02482025
Title: The Secure Messaging for Medication Reconciliation Tool (SMMRT) Trial
Acronym: SMMRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 14-059
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Drug-Related Side Effects and Adverse Reactions; Adverse Drug Events
Keywords: Medications; Hospitalization; Electronic medical records
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Usual care delivered at VA Boston
- SMMRT (Active Comparator): Receives Usual Care PLUS SMMRT Intervention
  Interventions: Other: SMMRT

INTERVENTIONS:
Other: SMMRT — Includes My HealtheVet registration and enrollment
  Arms: SMMRT

SUMMARY:
Medication discrepancies, defined as unintentional differences found between patients' medical records and patients' reports of the medication they are taking, occur frequently after hospital discharge, predisposing to adverse drug events (ADEs), emergency department visits and readmissions. Resolving medication discrepancies - medication reconciliation - is mandated at every care transition, but little is known about intervention strategies to improve medication reconciliation in the post-discharge period, when patients may lack prompt access to primary care and are at high risk for ADEs. To address this gap, the investigators developed and pilot tested the Secure Messaging for Medication Reconciliation Tool (SMMRT), with a pharmacist communicating with Veterans to review medications and reconcile discrepancies after hospital discharge via Secure Messaging (SM), within My HealtheVet (MHV), VA's patient portal. The objectives of The SMMRT Trial are therefore

To optimize the end-users' experience with SMMRT through usability testing and refinement of the tool; To conduct a randomized controlled trial (RCT) of usual care vs. usual care plus MHV Training vs. usual care plus MHV Training plus SMMRT to reduce hospital utilization; To evaluate how Veterans and staff perceived the impact of SMMRT on routine clinical practices and, specifically, on Veterans' interactions with their primary care providers.

DETAILED DESCRIPTION:
Study Procedure of Work Done at Richard L. Roudebush VAMC in Indianapolis

Aim 1 of SMMRT will be conducted at the Human-Computer Interaction & Simulation Laboratory within the HSR&D Center for Health Information and Communication at the Richard L. Roudebush VAMC in Indianapolis, IN. The work in Indianapolis will include a formal usability test of SMMRT to access and improve usability for pharmacists, nurses, and patients. Ten VA pharmacists, 10 VA nurses, and 10 VA patients will participate in the usability tests in Indianapolis. They will assess how well the SMMRT interface supports their respective medication reconciliation tasks. Pharmacists who work for the Roudebush VAMC and have some responsibility for medication reconciliation in their normal work will be eligible to participate in the study. Roudebush VAMC nurses who work as part of a Patient Aligned Care Team (PACT) will be eligible. Eligible patients must be taking at least 5 medications and must have been discharged from the Roudebush VAMC within the last 30 days. Veterans will be excluded if they are cognitively impaired, based on the Callahan screener. Patients will be recruited regardless of prior MHV use. No patients will have previous experience with SMMRT, as it is a new feature in MHV. Usability testing sessions will be about 30 minutes and will include audio and video recordings of the computer screen movements and the participant's face. A standardized script is read to the participants to instruct them to do certain tasks that will evaluate specific usability issues in the SMMRT. The participants enter reconciled medications into the SMMRT and the completed work is sent to the research team for analysis.

Although the investigators intend to complete all data collection procedures for Aim 1 at the Indianapolis VA, the investigators did note in the submitted grant proposal (Section 4.g.1) that the investigators would recruit (VA) Boston pharmacists for Aim 1 data collection in the unlikely event that the investigators cannot recruit sufficient numbers from Indianapolis. If that unlikely contingency arises (i.e., the investigators determine that there is a need to recruit pharmacists from VA Boston), the investigators will submit an amendment to the VA Boston IRB with appropriate consent and authorization forms at that time.

Study Procedure of Work at VABHS. The Study has received approval for a Project Modification.

The essential scientific changes of the proposed modification are (1) switching from a three-arm to a two-arm RCT; (2) changing the main outcome measure from hospital utilization to medication discrepancies; and (3) reducing the sample size from 1400 to 240 subject. The second specific aim of the Project will become the following:

Aim 2. To conduct a two-arm RCT to evaluate the effect of SMMRT. This trial will compare Usual Care (UC) with UC plus the bundled MHV/SMMRT Intervention among Veterans discharged from the VA Boston Community Living Center (CLC) and from the VA Boston acute inpatient setting of West Roxbury. The primary outcome measure will be medication discrepancies detected 30 days after discharge. Secondary outcome measures will be 30-day hospital utilization (combined readmissions plus emergency department use) and Veterans' self-efficacy in medication use. The primary hypothesis is that SMMRT will result in a reduction in 30-day medication discrepancies as compared with UC.

The third specific aim of the Project remains unchanged:

Aim 3. To evaluate the SMMRT intervention for potential future implementation. In anticipation of future implementation, we will use qualitative methods to identify features of the intervention that are most and least effective, as well as elements that are most and least likely to be accepted into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age 18 years or older
* Having a VA primary care provider (PCP) at any VA facility in VISN-1
* Planned discharge home (as opposed to another facility)
* Computer and internet access
* Anticipated to be discharged with at least 5 medications.

  * Having a VA PCP will be defined as having seen the provider within the past two years
  * Planned discharge home will be ascertained from the Veteran's nurse; approximately 75% of VA Boston discharges are to home
  * The nurse will also provide number of anticipated discharge medications

Exclusion Criteria:

* Cognitive impairment (as determined by the Callahan screener)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Linsky, MD MSc, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (1):
- VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Not sharing individual patient data.

REFERENCES:
- [Derived] Brady JE, Linsky AM, Simon SR, Yeksigian K, Rubin A, Zillich AJ, Russ-Jara AL. The Perceived Effectiveness of Secure Messaging for Medication Reconciliation During Transitions of Care: Semistructured Interviews With Patients. JMIR Hum Factors. 2022 Aug 3;9(3):e36652. doi: 10.2196/36652. PMID 35921139

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | SMMRT
Started | 122 | 118
Completed | 122 | 118
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Comparable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | SMMRT | Total
Number analyzed (Participants) | 122 | 118 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (11.8) | 63.4 (11.7) | 64.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 112 | 110 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 104 | 100 | 204
  Race: Non-White | 18 | 18 | 36
MyHealtheVet: Yes, No [Count of Participants; unit: Participants] — Was the Veteran already registered in My HealtheVet at the time of study enrollment? (Yes, No)
  Participants
    My HealtheVet - Yes | 107 | 105 | 212
    My HealtheVet - No | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Medication Discrepancies
Description: Medication discrepancies (discrepancies between what the patient is taking and what is in the medical record) identified 30 days after hospitalization via telephone interview and review of medical record
Time Frame: 30 days after hospitalization
Population: Intention to treat.
Measure: Mean (Standard Deviation); unit: Medication Discrepancies
Arm/Group | Usual Care | SMMRT
Number analyzed (Participants) | 122 | 118
Medication Discrepancies | 6.4 (4.6) | 4.4 (3.2)

2. Secondary Outcome: Hospital Utilization
Description: Hospital utilization, defined as re-admissions or emergency department utilization, within 30 days of hospital discharge.
Time Frame: 30 days
Population: Intention to Treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | SMMRT
Number analyzed (Participants) | 122 | 118
Participants | 41 | 35

ADVERSE EVENTS:
Time Frame: 30-day follow-up
Description: 30-day follow-up telephone calls
Arm/Group | Usual Care | SMMRT
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/118
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/118
Other Adverse Events (participants affected / at risk) | 0/122 | 0/118

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT02482025/Prot_SAP_000.pdf